CLINICAL TRIAL: NCT00003493
Title: Phase II Trial of Doxil, Vincristine and Decadron in Multiple Myeloma
Brief Title: Combination Chemotherapy in Treating Patients With Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CCF-IRB-2006; CDR0000066532 (Registry Identifier: PDQ (Physician Data Query)); SEQUUS-CCF-IRB-2006; NCI-V98-1459
Record Dates: First submitted 1999-11-01; First posted 2004-04-14 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2001-08

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: refractory multiple myeloma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Dexamethasone; Vincristine

INTERVENTIONS:
Drug: dexamethasone
Drug: pegylated liposomal doxorubicin hydrochloride
Drug: vincristine sulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy consisting of liposomal doxorubicin, vincristine, and dexamethasone in treating patients with newly diagnosed or previously treated multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the response rate and duration of response of multiple myeloma treated with doxorubicin HCl liposome, vincristine, and dexamethasone. II. Define the qualitative and quantitative toxic effects of this regimen in these patients.

OUTLINE: Patients are stratified into newly diagnosed (group A) and previously treated (group B) patients. Patients receive doxorubicin HCl liposome IV over 2.5 hours, followed by vincristine by bolus IV over 5 minutes on day 1. Dexamethasone is administered orally or by IV on days 1-4. Treatment is repeated every 4 weeks for a minimum of 6 courses, and 2 courses after maximum response unless unacceptable toxic effects or disease progression occur. Patients are followed until death.

PROJECTED ACCRUAL: A maximum of 33 patients from group A and 34 patients from group B will be accrued for this study within 6-14 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven newly diagnosed or previously treated multiple myeloma At least one chemotherapy regimen and no more than four regimens Pancytopenia related to multiple myeloma allowed At least 50% plasma cells in the bone marrow Splenomegaly OR Plasma cell leukemia No solitary bone or solitary extramedullary plasmacytoma

PATIENT CHARACTERISTICS: Age: Not specified Performance status: ECOG 0-2 Life expectancy: At least 3 months Hematopoietic: WBC at least 2,500/mm3 OR neutrophil count at least 1,000/mm3 (previously treated patients with platelet count at least 75,000/mm3 must have a neutrophil count of greater than 500/mm3) Platelet count at least 75,000/mm3 (previously treated patients must have platelet count at least 45,000/mm3) Thrombocytopenia related to idiopathic thrombocytopenic purpura or B12 or folate deficiency allowed Hepatic: Bilirubin no greater than upper limit of normal (ULN) ALT or AST no greater than 2 times ULN (unless greater than 1/3 of liver is involved by tumor, in which case ALT or AST must be no greater than 5 times ULN) Renal: Not specified Cardiovascular: LVEF at least 50% by MUGA scan or echocardiogram No New York Heart Association class II or greater cardiac disease Other: Not pregnant or nursing Fertile patients must use effective contraception No prior malignancies within 5 years, except: Adequately treated basal or squamous cell skin cancer Adequately treated carcinoma in situ of the cervix No uncontrollable physical, mental, or emotional disorders No history of hypersensitivity to doxorubicin HCL or liposomal or PEGylated formulations of other drugs No active infection requiring IV antibiotics

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Patients who have previously failed treatment with doxorubicin HCl liposome, vincristine, and dexamethasone (VAD) are allowed if anthracycline therapy has been at least 6 months, and prior anthracycline exposure no greater than 300 mg/m2 No other concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: Prior radiotherapy allowed Concurrent radiotherapy to control pain or prevent fractures allowed Surgery: Prior surgery allowed if recovered

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-11; Study Completion 2004-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad A. Hussein, MD, Study Chair — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio, United States